CLINICAL TRIAL: NCT06805266
Title: An Open Study to Evaluate the Efficacy of Vortioxetine on Freezing of Gait in Patients Affected by Parkinson Disease with Depressive Symptoms
Brief Title: Vortioxetine for Depressive Symptoms and Freezing of Gait in Parkinson Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Marianna Amboni (Other)
Responsible Party: Sponsor-Investigator, Marianna Amboni, Professor, University of Salerno
Organization: University of Salerno (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID:1279VTX - PD-20593T
Record Dates: First submitted 2025-01-16; First posted 2025-02-03 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease, Idiopathic; Freezing of Gait; Depression Not Otherwise Specified
Keywords: Parkinson Disease; freezing of gait; depression NOS
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Vortioxetine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FOG-PD (Experimental): FOG-PD will receive vortioxetine
  Interventions: Drug: Vortioxetine (tablet)

INTERVENTIONS:
Drug: Vortioxetine (tablet) — Vortioxetine will be used with the aim of treating freezing of gait in subjects with Parkinson Disease and depressive symptoms

SUMMARY:
The present study involves patients with Parkinson Disease (PD) suffering from freezing of gait (FOG) and depressive symptoms. The main aim of the study is evaluating the efficacy of vortioxetine in reducing moderate/severe FOG not responsive to dopaminergic treatment in patients with PD with depressive symptoms.

DETAILED DESCRIPTION:
Depression and anxiety are common in patients with Parkinson's disease (PD). In PD, several drugs, such as dopamine-agonists, inhibitors of serotonin uptake (SSRI), tricyclic antidepressants (TCAs) and norepinephrine uptake inhibitors (SNRI) are effective in treating depressive symptoms. Recently, a Delphi consensus has concluded that multimodal drugs, like vortioxetine, are good treatment options for depression in PD and an open-label prospective study has shown that the vortioxetine may improve depressive symptoms and cognition in PD patients with major depression Vortioxetine has different mechanisms of action; it is a serotonin transporter (SERT) inhibitor, an antagonist of 5-HT3, 5-HT7, 5-HTID, a partial agonist of 5-HT1B and a full agonist of 5-HT1A. Moreover, despite vortioxetine does not interact significantly with the norepinephrine transporters or dopamine transporters, it has been shown to increase extracellular levels of norepinephrine, dopamine, and non-monoamine neurotransmitters including acetylcholine. These effects are likely related to the interaction between vortioxetine and various serotonin receptors.

Depression and anxiety or panic attacks are commonly associated to freezing of gait (FOG) in PD. FOG is a disabling symptom of parkinsonian syndromes, whose pathophysiology is heterogeneous and partly unclear. The relationship between FOG and dopaminergic treatment is rather complex. Based on response to dopaminergic treatment, FOG may be responsive, unresponsive (or partially responsive) or induced by dopaminergic drugs. FOG, especially unresponsive FOG, is commonly associated with cognitive dysfunction, namely attentional-executive and visuospatial alterations in PD patients. Since FOG episodes might be related to the Off state and/or to dopaminergic underdosing in PD, the first treatment option should be the increase of dopaminergic drugs dose, when possible. FOG episodes that are less responsive or nonresponsive to dopaminergic treatment represent the greatest therapeutic challenge. Beyond dopaminergic pathway, non-dopaminergic networks, i.e. noradrenergic and cholinergic transmission, may play a role in the pathogenesis of FOG. We hypothesize that vortioxetine might be effective in treating FOG by enhancing both monoamine and non-monoamine neurotransmitters.

STUDY DESIGN Clinical evaluation will be performed during optimal on state of patients

VISIT 1:

1. Enrolment: Informed consent signature
2. Standardized gait analysis with wearable sensors:

   Patients will be videotaped and assessed with wearable sensors (Opal) while:

   A) Performing the Rating Instrument to Assess Festination and Freezing Gait in Parkinsonian Patients (RIAFFGPP) . In RIAFFGPP patients have to:

   i. Sit down on a chair set up in front of a door. ii. After 30 s, stand up and walk to a floor mark (40 x 40 cm) iii. Perform within the mark two 360° turns, clockwise (cw) and counter-clockwise (ccw) iiii. Open and walk through the door, turn outside, and come back to the chair

   B) Walking forward along a 10 m path during three conditions:

   i. self paced velocity ii. fastest as possible without running pace iii. self paced velocity with mental task (seven serial subtraction from 100 - counting aloud)
3. Clinical Global Impression scale (patient and clinician)
4. FOG Questionnaire referred to the on state
5. New freezing of gait questionnaire (NFOG-Q)
6. Falls Efficacy Scale
7. Cognitive function assessment:

   * MMSE
   * MoCA
   * FiPaT
   * Raven Progressive Matrices
   * The Benton Judgment of Line Orientation Test (JLOT)
   * Rey auditory 15-word learning test
   * Babcock story (episodic memory)
   * Rey Complex Figure (copy and recall)
   * Stroop test
   * Trial making test
   * Cancellation attentional matrices
   * Phonological verbal fluency
   * Semantic verbal fluency
   * Frontal Assessment Battery
   * Constructional Apraxia
   * SAND-Denomination
8. MDS-UPDRS
9. BDI-II
10. NPI
11. Apathy Scale
12. PDQ-8
13. Blood pressure, heart rate
14. Instruction to fill in a falls diary for the next 2 weeks

VISIT 2 (Start of treatment, after 14 days ± 3 days from Visit 1)

1. Enrolled patients will start vortioxetine:

   Vortioxetine Schedule:

   Vortioxetine 5 mg: once a day after lunch for one week, After one week, Vortioxetine 10 mg once a day
2. Instruction on filling in again a falls diary:

Four weeks after starting medication patients will fill in again a falls diary for the next 2 consecutive weeks

VISIT 3 (after 12 weeks ± 7 days from ):

1. Standardized gait analysis with wearable sensors (see visit 1)

   * RIAFFGPP
   * Walking forward along a 10 m path during three conditions
2. Clinical Global Impression scale (patient and clinician)
3. FOG Questionnaire
4. New freezing of gait questionnaire (NFOG-Q)
5. Falls Efficacy Scale
6. Cognitive function assessment (see visit 1)
7. MDS-UPDRS or
8. BDI-II
9. NPI
10. Apathy Scale
11. PDQ-8
12. Blood pressure, heart rate
13. Adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PD according to published criteria
2. Occurrence of depression according to Beck Depression Inventory II (score ≥ 15)
3. A score ≥ 2 on the freezing question #2.13 of part 2 of the MDS-UPDRS (moderate-severe FOG).
4. FOG not responsive to dopaminergic treatment.

Exclusion Criteria:

1. Treatment with IMAO-B (rasagiline, selegiline, safinamide) (to be included, IMAO-B need to be withdrawn for at least 15 days)
2. Concomitant treatment with other antidepressant drugs
3. Hepatic and renal insufficiency
4. Treatment with tramadol or triptans
5. Psychotic disorder
6. Dementia according to DSM-V

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in the score of the Freezing Of Gait (FOG) Questionnaire referred to the "on state" | From enrollment to the end of treatment at 12 weeks
  Total score of FOG Questionnaire ranges from 0 to 24 and higher scores correspond to more severe FOG

SECONDARY OUTCOMES:
Change on severity of FOG not responsive to dopaminergic treatment in patients with PD. | From enrollment to the end of treatment at 12 weeks
  Change on duration (seconds) of FOG episodes on standardized gait analysis with wearable sensors
Chenage on frequency of FOG not responsive to dopaminergic treatment in patients with PD. | From enrollment to the end of treatment at 12 weeks
  Change on number of FOG episodes on standardized gait analysis with wearable sensors

IPD SHARING:
Plan to Share IPD: Yes
Clinical and outcome measures
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For 12 months after the completation of the study
Access Criteria: contacting Central Contact Person by email on mamboni@unisa.it

REFERENCES:
- [Background] Ziegler K, Schroeteler F, Ceballos-Baumann AO, Fietzek UM. A new rating instrument to assess festination and freezing gait in Parkinsonian patients. Mov Disord. 2010 Jun 15;25(8):1012-8. doi: 10.1002/mds.22993. PMID 20310009
- [Background] Santos Garcia D, Alonso Losada MG, Cimas Hernando I, Cabo Lopez I, Yanez Bana R, Alonso Redondo R, Paz Gonzalez JM, Cores Bartolome C, Feal Painceiras MJ, Iniguez Alvarado MC, Labandeira C, Garcia Diaz I. Vortioxetine Improves Depressive Symptoms and Cognition in Parkinson's Disease Patients with Major Depression: An Open-Label Prospective Study. Brain Sci. 2022 Oct 29;12(11):1466. doi: 10.3390/brainsci12111466. PMID 36358393
- [Background] Nieuwboer A, Rochester L, Herman T, Vandenberghe W, Emil GE, Thomaes T, Giladi N. Reliability of the new freezing of gait questionnaire: agreement between patients with Parkinson's disease and their carers. Gait Posture. 2009 Nov;30(4):459-63. doi: 10.1016/j.gaitpost.2009.07.108. Epub 2009 Aug 5. PMID 19660949
- [Background] Bloem BR, Marinus J, Almeida Q, Dibble L, Nieuwboer A, Post B, Ruzicka E, Goetz C, Stebbins G, Martinez-Martin P, Schrag A; Movement Disorders Society Rating Scales Committee. Measurement instruments to assess posture, gait, and balance in Parkinson's disease: Critique and recommendations. Mov Disord. 2016 Sep;31(9):1342-55. doi: 10.1002/mds.26572. Epub 2016 Mar 4. PMID 26945525
- [Background] Bang-Andersen B, Ruhland T, Jorgensen M, Smith G, Frederiksen K, Jensen KG, Zhong H, Nielsen SM, Hogg S, Mork A, Stensbol TB. Discovery of 1-[2-(2,4-dimethylphenylsulfanyl)phenyl]piperazine (Lu AA21004): a novel multimodal compound for the treatment of major depressive disorder. J Med Chem. 2011 May 12;54(9):3206-21. doi: 10.1021/jm101459g. Epub 2011 Apr 12. PMID 21486038
- [Background] Amboni M, Stocchi F, Abbruzzese G, Morgante L, Onofrj M, Ruggieri S, Tinazzi M, Zappia M, Attar M, Colombo D, Simoni L, Ori A, Barone P, Antonini A; DEEP Study Group. Prevalence and associated features of self-reported freezing of gait in Parkinson disease: The DEEP FOG study. Parkinsonism Relat Disord. 2015 Jun;21(6):644-9. doi: 10.1016/j.parkreldis.2015.03.028. Epub 2015 Apr 13. PMID 25899545
- [Background] Amboni M, Cozzolino A, Longo K, Picillo M, Barone P. Freezing of gait and executive functions in patients with Parkinson's disease. Mov Disord. 2008 Feb 15;23(3):395-400. doi: 10.1002/mds.21850. PMID 18067193
- [Background] Aguera-Ortiz L, Garcia-Ramos R, Grandas Perez FJ, Lopez-Alvarez J, Montes Rodriguez JM, Olazaran Rodriguez FJ, Olivera Pueyo J, Pelegrin Valero C, Porta-Etessam J. Focus on Depression in Parkinson's Disease: A Delphi Consensus of Experts in Psychiatry, Neurology, and Geriatrics. Parkinsons Dis. 2021 Feb 8;2021:6621991. doi: 10.1155/2021/6621991. eCollection 2021. PMID 33628415